CLINICAL TRIAL: NCT02245256
Title: Perioperative Low-dose Dexmedetomidine Decreases Incidence of Delirium in Liver Transplant Patients
Brief Title: Efficacy of Low-dose Dexmedetomidine to Prevent Delirium in Liver Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Ho Geol Ryu, assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1407-114-596
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Liver Transplantation
Keywords: delirium; incidence; dexmedetomidine
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal saline (Placebo Comparator): same infusion rate as experimental group (dexmedetomidine)
  Interventions: Drug: placebo control
- dexmedetomidine (Experimental): 0.1mcg/kg/hr of dexmedetomidine infusion started after induction of anesthesia for liver transplantation and continued until 48 hours after surgery.
  Interventions: Drug: Precedex

INTERVENTIONS:
Drug: Precedex — infusion of 0.1mcg/kg/hr of precedex
  Arms: dexmedetomidine
Drug: placebo control — placebo
  Other Names: 0.9% saline
  Arms: Normal saline

SUMMARY:
To test the effect of low-dose dexmedetomidine for lowering the incidence of postoperative delirium in liver transplant patients in the ICU.

Single center prospective randomized placebo controlled clinical trial 0.1mcg/kg/hr of dexmedetomidine or equivalent amount of saline infusion started after induction of anesthesia for liver transplantation and continued until 48 hours after surgery.

Outcomes will be assessed up to 1 week or transfer to ward, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18years old or older) undergoing living-donor or deceased-donor liver transplantation

Exclusion Criteria:

* Pediatric patients (under 18 years) Pregnancy Patients who are unresponsive at baseline, who have neurologic deficits at baseline, or who are allergic to dexmedetomidine

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
analysis of the incidence of postoperative delirium in liver transplant patients in the ICU. | 1 week or transfer to ward, whichever comes first.
  after August 25, 2014

SECONDARY OUTCOMES:
analysis of the duration of postoperative delirium, ICU length of stay in liver transplant patients in the ICU. | 1 week or transfer to ward, whichever comes first.
  after August 26, 2014

CONTACTS AND LOCATIONS:
Overall Officials: Hogeol Ryu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Agree, South Korea

REFERENCES:
- See also: Related Info — http://www.icudelirium.org